CLINICAL TRIAL: NCT06662773
Title: Phase I Clinical Trial Evaluating Drug Drug Interactions of TQB3616 Capsules
Brief Title: Drug-Drug Interaction (DDI) Study for TQB3616
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-I-05
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitor group (Experimental): Oral TQB3616 capsules 60 mg after a single meal on days 1 and 13; On days 10 to 21, itraconazole capsules 200mg were taken orally once a day for 12 days after meals.
  Interventions: Drug: TQB3616 capsule + itraconazole
- Inducer group (Experimental): 180mg of TQB3616 capsules orally after a single meal on days 1 and 17; Oral administration of rifampicin capsules 600mg from day 10 to day 25 on the peritoneum once a day for 16 consecutive days, of which rifampicin capsules 600mg and TQB3616 capsules 180mg were taken at the same time after meals on the 17th day.
  Interventions: Drug: TQB3616 capsule + rifampicin

INTERVENTIONS:
Drug: TQB3616 capsule + itraconazole — C2/4/6 inhibitors + CYP3A metabolic enzyme inhibitors
  Arms: Inhibitor group
Drug: TQB3616 capsule + rifampicin — C2/4/6 inhibitors + Non-specific cytochrome P450 enzyme inducer
  Arms: Inducer group

SUMMARY:
To evaluate the effect of itraconazole/rifampicin on the pharmacokinetics of TQB3616 capsules.

To assess the safety of a single dose of oral TQB3616 capsules and in combination with itraconazole/rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form, the age is 18~45 years old (including the cut-off value), both male and female;
* Females ≥ 45kg, males ≥ 50kg, body mass index (BMI) is 19~26 kg/m^2 (including the critical value), BMI = weight (kg)/height^2 (m^2);
* Those with normal vital signs, physical examination, clinical laboratory examination, imaging examination, 12-lead electrocardiogram, or abnormal but no clinical significance as judged by the investigator;
* Subject is able to comply with study procedures, voluntarily participate in this trial, and sign an informed consent form in writing.

Exclusion Criteria:

* Those who have suffered or are currently suffering from any clinically serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematology, immunology, psychiatry and metabolic abnormalities or any other diseases that can interfere with the test results;
* Those who have systemic/local acute infection before taking the study drug;
* Those with a history of food or drug allergies, or allergies;
* Those who have dysphagia or suffer from any gastrointestinal diseases that affect drug absorption at the time of screening;
* Those who cannot accept intravenous indwelling needle puncture blood vessels to collect blood samples, or the subjects cannot tolerate venipuncture, or have a history of needle fainting or blood sickness;
* Regular drinkers within 6 months before the first dose, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine) or those who have a positive alcohol breath test at screening;
* History of major surgical operation (defined as difficult and complex intraoperative surgery, such as gastric and duodenal surgery, partial nephrectomy, radical resection of malignant tumor, etc.) within 3 months before the first dose, or have taken investigational drugs or participated in other drug clinical trials;
* Blood donation or massive blood loss (>400 mL) within 3 months before the first dose;
* Those who have used drugs within 3 months before the first dose, or those who have a positive drug screen, or those who have a history of drug abuse within five years before screening;
* Those who smoke more than 5 cigarettes per day within 3 months before the first dose or those who cannot stop using any tobacco products during the trial;
* Daily consumption of excessive tea, coffee, and/or caffeinated beverages (more than 8 cups, 1 cup=250 mL) within 30 days prior to the first dose;
* Use of any drug that inhibits or induces the hepatic metabolism of the drug within 30 days before the first dose (such as: CYP3A4 inducers carbamazepine, dexamethasone, rifampicin, phenytoin, phenobarbital, St. John's worn, etc.); CYP3A4 inhibitors itraconazole, ketoconazole, clarithromycin, telithromycin, lopinavir, ritonavir, etc.);
* Have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 14 days before the first dose;
* Those who have taken a special diet (such as grapefruit) or other factors that affect the absorption, distribution, metabolism, and excretion of drugs within 7 days before the first dose;
* Ingestion of chocolate, any caffeine-containing, or xanthine-rich food or drink 48 hours prior to the first dose;
* Those who have special dietary requirements and cannot comply with the unified diet;
* Pregnant or lactating women, as well as subjects and their spouses who have childbearing, or sperm donation, or egg donation plans within 3 months from signing the informed consent form to the last dose, or who cannot guarantee the use of effective contraception during this period (taking one or more non-drug contraceptive measures during the trial);
* Subjects who are judged by the investigator to be unsuitable to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Before administration, 1,2,4,6,8,12,24,48,72,120,168,216 hours after administration
  Maximum plasma drug concentration
Area under drug time curve (AUC0-t) | Before administration, 1,2,4,6,8,12,24,48,72,120,168,216 hours after administration
  Area under the plasma concentration time curve from time 0 to last time of quantifiable concentration.
Area under drug time curve (AUC0-∞) | Before administration, 1,2,4,6,8,12,24,48,72,120,168,216 hours after administration
  Area under the plasma concentration-time curve from time 0 extrapolated to infinite time.

SECONDARY OUTCOMES:
Adverse event rate | From before the first administration to 26 days after the administration
  Incidence and severity of adverse events and serious adverse events, and abnormal laboratory examination indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China